CLINICAL TRIAL: NCT07139431
Title: A Study to Evaluate the Cellular Distribution of [89Zr]-Oxine-NCR100 Injection in the Treatment of Subjects With Knee Osteoarthritis
Brief Title: A Study of [89Zr]-Oxine-NCR100 Injection for the Cellular Distribution
Acronym: Distribution
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCR100-1003
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: KOA
Keywords: MSC, KOA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCR100 injection (Experimental): Subjects will receive a single injection of NCR100
  Interventions: Biological: NCR100

INTERVENTIONS:
Biological: NCR100 — Subjects will receive a single injection of NCR100

SUMMARY:
This clinical study is to evaluate the biodistribution of [89Zr]-Oxine-NCR100 injection in subjects with knee osteoarthritis after local injection and the kinetic behavior characteristics of zirconium-labeled cells at the injection site and various organs or tissues. It is a single-dose, open-label study in adult KOA subjects.

DETAILED DESCRIPTION:
Knee osteoarthritis(KOA) is a kind of degenerative joint disease characterized by chronic inflammation loss of articular cartilage and subchondral bone remodeling. This clinical trial aims to evaluate the biodistribution of 89Zr-labeled human pluripotent stem cell derived mesenchymal stromal cells ([89Zr]-Oxine-NCR100) injection in subjects with knee osteoarthritis after local injection and the kinetic behavior characteristics of the zirconium-labeled cells at the injection site and in various organs or tissues.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and voluntarily sign the Informed Consent Form（ICF） before enrolment; Age: 40-70 years old, both genders; Men without reproductive intentions; Diagnosis of knee osteoarthritis based on American College of Rheumatology criteria.

Subjects with KOA who have persistent pain for more than six months, Kellgren-Lawrence grade: II-III; McMaster University's Osteoarthritis Index (WOMAC) of the study-side knee joint: 60-180.

Exclusion Criteria:

* Subjects previously diagnosed with secondary knee osteoarthritis, or those diagnosed with hip/ankle joint disease requiring medical intervention; Subjects previously diagnosed with secondary knee osteoarthritis, or those diagnosed with hip/ankle joint disease requiring medical intervention; Have received stem cell therapy; Experienced knee surgery, or plan to undergo knee surgery; Have used traditional Chinese medicine to treat KOA within 4 weeks; Have used intra-articular injection of drugs to treat KOA within 12 weeks; Received glucosamine, chondroitin sulfate, or diacetate therapy before investigational drug intervention within 12 weeks; Subjects with the acute phase of knee osteoarthritis; severe deformity of the knee; BMI≥30kg/m^2; Severe systemic infection or local knee joint infection; Have received systemic glucocorticoid therapy before intervention or need to take systemic glucocorticoid therapy during the treatment; Have serious heart disease； Subjects with peripheral or central nervous system disorders that may interfere with assessments; Have contraindications to Magnetic Resonance Imaging(MRI); Subjects with alcohol/drug addiction/abuse or mental disorders; Have participated in other clinical trials within 12 weeks before the screening; Subjects with infection with hepatitis B virus(HBV), hepatitis C virus(HCV), HIV, and Treponema pallidum confirmed by laboratory tests; Subjects with a history of allergic reaction to any component of the trial drug or to acetaminophen; Subjects who are not suitable for PET/CT examination.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2026-03-06 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
The Standardized Uptake Values (SUV) and %ID | Day2, Day8,Day12,and Day22
  The SUV and %ID of the injection site and various organs or tissues after PET/CT imaging examination after local injection of [89Zr]-Oxine-NCR100 injection in subjects with knee osteoarthritis

SECONDARY OUTCOMES:
Adverse Event(AE) or Serious Adverse Event(SAE) | Within 96 weeks of the infusion
  Number of participants with treatment-related adverse events or serious adverse events assessed by CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No